CLINICAL TRIAL: NCT03516578
Title: Comprehensive Cardiac Magnetic Resonance Imaging For Prognosis Assessment After Non-ST-Elevation Myocardial Infarction
Brief Title: CMR for Prognosis Assessment in NSTEMI
Status: Completed | Type: Observational
Sponsor: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1
Record Dates: First submitted 2018-04-24; First posted 2018-05-04 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Myocardial Infarction
Keywords: non-ST-elevation myocardial infarction; cardiac magnetic resonance; prognosis
MeSH Terms: conditions — Myocardial Infarction; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Cardiac magnetic resonance imaging

SUMMARY:
The prognostic significance of cardiac magnetic resonance (CMR) derived parameters of myocardial and microvascular injury has not been fully elucidated yet in non-ST-Elevation myocardial infarction (NSTEMI) patients. In the present study the investigators aim to comprehensively investigate the prognostic significance of CMR in a prospective, multicentre registry cohort of NSTEMI patients undergoing early percutaneous coronary intervention (PCI). CMR will be performed within the first week following the index event. The primary endpoint is defined as a composite of death, reinfarction, and new congestive heart failure (major adverse cardiac events) at 12 months.

ELIGIBILITY:
Inclusion Criteria: Patients are eligible for the study if they have: 1) ischemic symptoms in accordance with a possible NSTEMI diagnosis; 2) elevated cardiac troponin levels above the 99th percentile; and 3) identifiable culprit lesion during early invasive coronary angiography with performed PCI.

Exclusion Criteria: 1) STEMI; 2) presence of cardiogenic shock; 3) no identifiable culprit lesion or culprit lesion ineligible for PCI; 4) indication for acute bypass surgery; 5) age less than 18 years or more than 90 years; 6) pregnancy; and 7) typical contraindications to CMR (e.g. severe claustrophobia, implanted pacemakers and internal cardioverter defibrillators, cerebral or intracranial metallic implants, known allergy to gadolinium and creatinine clearance <30 mL/min).

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the chest pain units of three primary care clinics are screened for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2018-03-28 (Actual); Study Completion 2018-03-28 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac events | 12 months
  Composite of death, reinfarction and new congestive heart failure

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Feistritzer HJ, Nanos M, Eitel I, Jobs A, de Waha-Thiele S, Meyer-Saraei R, Freund A, Stiermaier T, Abdel-Wahab M, Lurz P, Reinstadler SJ, Reindl M, Klug G, Metzler B, Desch S, Thiele H. Determinants and prognostic value of cardiac magnetic resonance imaging-derived infarct characteristics in non-ST-elevation myocardial infarction. Eur Heart J Cardiovasc Imaging. 2020 Jan 1;21(1):67-76. doi: 10.1093/ehjci/jez165. PMID 31518417
- [Derived] Feistritzer HJ, Eitel I, Jobs A, de Waha-Thiele S, Stiermaier T, Abdel-Wahab M, Lurz P, Reinstadler SJ, Reindl M, Klug G, Metzler B, Desch S, Thiele H. Impact of smoking on cardiac magnetic resonance infarct characteristics and clinical outcome in patients with non-ST-elevation myocardial infarction. Int J Cardiovasc Imaging. 2019 Jun;35(6):1079-1087. doi: 10.1007/s10554-019-01556-2. Epub 2019 Feb 15. PMID 30771036